UCD0115B: An Open-label Extension Study of Purified Epicatechin to Improve Mitochondrial Function, Strength and Skeletal Muscle Exercise Response in Becker Muscular Dystrophy

NCT03236662

**August 20, 2015** 


*Title of research study:* UCD0115B: An open-label extension study of purified epicatechin to improve mitochondrial function, strength and skeletal muscle exercise reponse in Becker Muscular Dystrophy.

Investigator: Craig McDonald, MD

## Why am I being invited to take part in a research study?

We invite you to take part in this extension research study because you are an adult diagnosed with Becker muscular dystrophy and were previously enrolled in the Pilot Epicatechin study.

#### What should I know about a research study?

(Experimental Subject's Bill of Rights)

- Someone will explain this research study to you, including:
  - o The nature and purpose of the research study.
  - o The procedures to be followed.
  - Any drug or device to be used.
  - Any common or important discomforts and risks.
  - Any benefits you might expect.
  - Other procedures, drugs, or devices that might be helpful, and their risks and benefits compared to this study.
  - Medical treatment, if any, that is available for complications.
- Whether or not you take part is up to you.
- You can choose without force, fraud, deceit, duress, coercion, or undue influence.
- You can choose not to take part.
- You can agree to take part now and later change your mind.
- Whatever you decide it will not be held against you.
- You can ask all the questions you want before you decide.
- If you agree to take part, you will be given a signed and dated copy of this document.
- If you agree to take part, you will be given a copy of this document.

#### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team:

| Craig McDonald, MD | Study PI | _at phone number <u>916-734-2923</u> |
|---|---|---|
| Erik Henricson, MPH | Co-PI | _at phone number <u>916-734-5294</u> |
| Candace Aguilar | Study Coordinator | _at phone number <u>916-734-0968</u> |

UC Davis Department of Physical Medicine and Rehabilitation 4860 Y Street, Suite 3850 Sacramento, CA 95817

For emergencies please call the following 24-hour emergency number. Our study doctors are available 24 hour a day for these health related emergencies.

#### UC Davis Medical Center operator - (916) 734-2011 (Ask for the PM&R Resident on call)

This research has been reviewed and approved by an Institutional Review Board ("IRB"). Information to help you understand research is on-line at <a href="http://www.research.ucdavis.edu/policiescompliance/irb-admin/">http://www.research.ucdavis.edu/policiescompliance/irb-admin/</a>. You may talk to a IRB staff member at (916) 703-9151, <a href="https://www.research.ucdavis.edu/policiescompliance/irb-admin/">IRBAdmin@ucdmc.ucdavis.edu/</a>, or 2921 Stockton Blvd, Suite 1400, Room 1429, Sacramento, CA 95817 for any of the following:

| | nstitutional Review Board<br>of California, Davis |
|----------|---------------------------------------------------|
| Protocol | Approved |
| 767161 | 08/20/2015 |


- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

#### Why is this research being done?

This research study will test an investigational drug called (-)-Epicatechin. New drugs or biologics that have not yet been approved by the FDA or approved drugs that have not yet been approved for a new use, and are in the process of being tested for safety and effectiveness. (-)-Epicatechin is purified from tea as a nutritional extract. (-)-Epicatechin will be evaluated for the treatment of progressive muscle loss and impaired skeletal muscle function in Becker Muscular Dystrophy (BMD) patients.

(-)-Epicatechin has been shown to improve muscle structure and function in previous studies of animals and humans. This study drug is not currently approced by the Food and Drug Administration (FDA) for the treatment of BMD.

The main objective of this study is to test your blood samples for biomarkers and determine whether or not the study drug is affecting these molecules and possibly the structure and function of you muscles.

#### How long will the research last?

We expect that you will be in this research study for 48 weeks for a total of 8 visits. Each visit on average will be expected to be about a 3 hours induration.

## How many people will be studied?

We expect about 10 people here will be in this research study at UC Davis.

#### What happens if I say yes, I want to be in this research?

#### **Study Procedures:**

See below for a table of all the study procedures

| Event | Screening | Baseline | PK Week 4 | Week 8 | Week 12 | Week 24 | Week 36 | Week 48 |
|---|---|---|---|---|---|---|---|---|
| | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 |
| | Day -28 to 0 | Day 1 | Day 28 | Days 53-<br>59 | Days 81-87 | Days 165-171 | Days 249-255 | Days 333-339 |
| Informed consent | Х | | | | | | | |
| Medical history | Х | Х | Х | Х | Х | Х | Х | Х |
| Vital signs | Х | Х | Х | Х | Х | Х | Х | Х |
| Physical examination | Х | Х | Х | Х | Х | Х | Х | Х |
| Adverse Event/<br>Medications | Х | Х | | Х | Х | х | х | х |
| ECG | Х | Х | Х | Х | Х | | Х | Х |
| PK | | Pre, 2H, 4H | Pre | | Pre | Pre | Pre | Pre |

| For IRB Us | se | |
|------------|----------|-----------------------------------------------------|
| | • | Institutional Review Board ity of California, Davis |
| | Protocol | Approved |
| | 767161 | 08/20/2015 |
| i | • | |


| Complete Blood<br>Count/Serum<br>Chemistries/Urinalysis | × | | x | х | х | х | x | х |
|---|---|---|---|---|---|---|---|---|
| Tbsp. of Blood Volume | 7 tbsp. | 4 tbsp. | 8 tbsp. | 6 tbsp. | 9 tbsp. | 9 tbsp. | 9 tbsp. | 9 tbsp. |
| Fasting Insulin, Glucose | Х | | | | Х | × | × | х |
| Biomarkers | | Х | Х | | Х | Х | Х | Х |
| Functional assessments | | Х | × | | X | x | × | х |
| DEXA | | Х | Х | | Х | Х | Х | Х |
| Dispense Epicatechin | Х | Х | Х | X | Х | Х | Х | Х |
| Questionnaire | Х | | | X | | | | |

<sup>\*</sup>Multiple blood draws at visits 2, 3, 5, 6, 7, 8.

## Informed consent (30 mins) (At Screening)

Before we begin any procedure we will review this consent form with you and answer any questions that you might have. After you sign the consent form we will provide you with a copy.

#### Medical history

We will ask you questions about medical conditions

#### Vital signs and physical exam

We will measure your weight, height, blood pressure and breathing rate.

#### Adverse events/ Medications

We will ask you about medications that you are taking and if anything has happened since the last visit that hurt or was out of the ordinary with regard to your health.

#### Safety & Drug monitoring/ blood & urine collection

During each visit we will perform blood draw(s) and one urine sample collection for safety assessments.

We will collect the following blood samples:

- Complete blood count/Serum chemistries- 6 tablespoons/18 teaspoons
- Biomarker- 1 tablespoon/3 teaspoons
- Fasting insulin/glucose- 1 tablespoon/3 teaspoons
- PK (protein kinase)- 1 tablespoon/3 teaspoons

#### Electrocardiogram (ECG)

This test will provide information on how well your heart is working. .

#### Strength & Exercise Testing

You will be asked to perform several exercise tests including the following measures:

| | nstitutional Review Board<br>of California, Davis |
|----------|---------------------------------------------------|
| Protocol | Approved |
| 767161 | 08/20/2015 |


- Six minute walk test—you will walk as fast as you can for 6 minutes around 2 cones
- Recumbent cycling test—you will exercise using a recumbent bicycle
- Assisted six minute cycle test---you will cycle as fast as you can for 6 minutes
- Strength test—we will measure the strength of your elbows and knees with a BIODEX ergometer (hand and arm operated bicycle)
- Range of motion test—we will assess your range of motion by measuring the extension of your knees, ankles, elbows and wrists in front of a motion sensing system
- Breathing tests—you will perform PFTs (Pulmonary Function Tests) to assess how much air you can breathe in and out
- Timed Function Testing—we will assess your ability to rise from the floor, climb four standard stairs and walk or run for 10 meters
- Upper/Lower Extremity function—we will assess your ability to use your arms and legs
- Anthropometric Measurements—we will measure your waist and hip circumference
- Body Composition by Dual energy X-ray absorptiometry (DEXA)—we will ask you to lie still on
  the bed of the DEXA scanner. The scanning arm will pass over your body one or more times
  and will make a computerized X-ray image of your whole body. You will not feel anything during
  the scan, but you will be asked to lie very still. The purpose of adding this measure to our study
  is to find out your body composition.
- Multifrequency Bioimpedence Assessment (MFBIA)—we will assess the amount of total water and fat-free mass in your body. Electrodes are placed on your ankle and wrist. Impedence is measured between upper and lower extremity electrodes. You will not feel anything during the test.

#### Study Medication-Epicatechin

- Medications will be dispensed for the entire period of time between study. The site will dispense
  study medication to you and you will keep a medication log to document all study medication
  dispensed. You will be instructed to take the study medication per dosing schedule, every day
  during the eight-week treatment period. You will be asked to return your empty medication
  container and/or any remaining pills at the next visit.
- You will swallow pills of (-)-epicatechin 50mg twice per day (100mg per day total dose). Study medication will be supplied as a clear 25mg gelatin capsule. You will take two capsules in the morning at approximately 7:30AM at least 15 minutes before the morning meal and two with the evening at approximately 7:30PM at least 1 hour after the evening meal.

#### What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible to: Tell the doctor if you have any new or worsening medical symptoms or problems during the time you receive the study medication as part of this study. It is important that you tell the doctor even if symptoms or problems are mild or you do not think they are related to study drug.

You will need to complete a drug diary and bring your medication to each study visit.

Please call if you have any questions about study medication or about the use of other drugs during the time that you receive study medication.

| | nstitutional Review Board<br>of California, Davis |
|----------|---------------------------------------------------|
| Protocol | Approved |
| 767161 | 08/20/2015 |


Contact the doctor immediately if an overdose of study drug happens or is suspected.

#### What happens if I do not want to be in this research?

You may decide not to take part in the research and it will not be held against you as participation is on a voluntary basis.

Instead of being in this research study, your choices may include: participating in other available clinical trials or choosing not to participate at all.

#### What happens if I say yes, but I change my mind later?

You can leave the research at any time and it will not be held against you.

If you decide to leave the research, contact the investigator so that the investigator can can recommend proper follow up care.

If you stop being in the research, already collected data may not be removed from the study database. You will be asked whether the investigator can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

#### Is there any way being in this study could be bad for me?

#### **Potential Risks**

#### Risks of Study Medication (Epicatechin)

Hypotension (low blood pressure). Given the reported effects of (-)-epicatechin on blood vessels, it a potential risk may be associated with hypotension. With cocoa based studies, blood pressure reducing effects are only reported in humans that have high blood pressure. There is the possibility that patients undergoing drug treatment for high blood pressure if given (-)-epicatechin may develop hypotension.

*Migraines (Headaches).* The consumption of cocoa products has been associated with increased likelihood of migraine development. (-)-Epicatechin may increase the chances for migraine development in certain individuals.

*Bleeding*. Anti-clotting like effects have been described in a limited number of reports on the effects of cocoa, although no such reactions have been seen to date. It will be important not to take any "blood thinning" medications (example: Asprin and Advil) during the study without consulting the study doctor.

#### Risks of Blood Tests

The risks of blood drawing include soreness or bruising at the site of the needle. A local numbing cream (EMLA) may be applied to the area. There are no side effects associated with the use of this cream. Rarely, a more serious injury, such as hematoma (bleeding under skin) or infection may develop. Repeated blood draw may increase the chance of the risks above.

#### Risks of Strength Testing and Functional Assessments

At this time, there are no known risks associated with functional evaluation or muscle strength testing methods used in this protocol. However, you may experience mild muscle soreness the day after muscle testing.

#### Risks of Breathing Tests

These tests may cause dizziness and lightheadedness during and shortly after the test.

#### Risks of Electrocardiogram (ECG)

| | nstitutional Review Board<br>of California, Davis |
|----------|---------------------------------------------------|
| Protocol | Approved |
| 767161 | 08/20/2015 |


The ECG has no known risks.

#### Risks of DEXA

This study involves a low radiation exposure that is less than other diagnostic tests using ionizing radiation. The amount of radiation exposure received in this study is below the levels that are thought to result in a significant risk of harmful effects.

## Risks of Multi-Frequency Bioimpedence Assessment (MFBIA)

There are no known risks of MFBIA testing.

#### Risks of Upper Extremity Range of Motion Evaluation

There are no known risks of upper extremity range of motion evaluation.

#### Risk of Pregnancy

The research may also hurt a pregnancy or fetus in ways that are unknown. The subject should not father a baby while in this study, and they should not donate semen/sperm or have vaginal sex (intercourse) without using effective birth control.

## Will being in this study help me in any way?

It is possible the participants will not experience any direct benefit as a result of their study participation. However, the data collected during this trial may provide information that will benefit the scientific community as well as other individuals with BMD

#### What happens to the information collected for the research?

Efforts will be made to limit use or disclosure of your personal information, including research study and medical records, to people who have a need to review this information. We cannot promise complete confidentiality. Organizations that may inspect and copy your information include the IRB and other University of California representatives responsible for the management or oversight of this study.

The IRB and the Food and Drug Administration will be granted direct access to your research records to conduct and oversee the study. We may publish the results of this research. However, we will keep your name and other identifying information confidential.

During your participation in this research, data will be collected about you. The de-identified data and any specimens, such as blood or tissue, are taken from you for this study, they will become the property of the University of California. The specimens may be used in this research, may be used in other research, and may be shared with other organizations. The specimens could lead to discoveries or inventions that may be of value to the University of California or to other organizations. Under state law you do not have any right to money or other compensation stemming from products that may be developed from the specimens.

If you agree to share the biological specimen(s) collected from you, please initial here.

Otherwise, your specimen will be destroyed at the end of this study. Information regarding biomarkers and outcome of the study will not be shared.

The sponsor, monitors, auditors, the IRB, the Food and Drug Administration will be granted direct access to your research records to conduct and oversee the study. We may publish the results of this research. However, we will keep your name and other identifying information confidential.

| | nstitutional Review Board of California, Davis |
|----------|------------------------------------------------|
| Protocol | Approved |
| 767161 | 08/20/2015 |


A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

If we access protected health information (e.g., your medical record), you will be asked to sign a separate form to give your permission. Your medical records may become part of the research record. If that happens, your research records may be looked at by the sponsor of this study and government agencies or other groups associated with the study. They may not copy or take your personal health information from your medical records unless permitted or required by law.

Federal law provides additional protections of your medical records and related health information. These are described in the UC Davis Health System Notice of Privacy Practices (<a href="http://www.ucdmc.ucdavis.edu/compliance/pdf/notice.pdf">http://www.ucdmc.ucdavis.edu/compliance/pdf/notice.pdf</a>) and in an attached document.

#### Can I be removed from the research without my OK?

. The person in charge of the research can remove you from the research study without your approval in circumstances when new information regarding safety in this trisl or other trials involving new safety concerns with Epicatechin. We will tell you about any new information that may affect your health, welfare, or choice to stay in the research

#### What else do I need to know?

There is no charge for you to participate in this study. Neither you nor your insurance carrier will be charged for your taking part in the research. All costs associated with the study will be paid by the sponsor/department.

It is important that you promptly tell the person in charge of the research if you believe that you have been injured because of taking part in this study. If you are injured as a result of being in this study, the University of California will provide necessary medical treatment. Depending on the circumstances, the costs of the treatment may be covered by University or the study sponsor or may be billed to your insurance company just like other medical costs. The University does not normally provide any other form of compensation for injury.

You will not be compensated for taking part in this study.

For more information about compensation, you may call the IRB Administration at (916) 703-9151 or email at IRBAdmin@ucdmc.ucdavis.edu.

| Your signature documents your permission to take part in this research | ch. |
|---|---|
| Signature of subject | Date |
| Printed name of subject | |
| Signature of person obtaining consent | Date |

| For IRB U | se | |
|-----------|----------|-----------------------------------------------------|
| | | nstitutional Review Board<br>y of California, Davis |
| | Protocol | Approved |
| | 767161 | 08/20/2015 |
| i | | |

| | |
|---|---|
| Printed name of person obtaining consent Signature Block for Capable Adult | |
| My signature below documents that the information in the consent documents information was accurately explained to, and apparently understood by, was freely given by the subject. | |
| Signature of witness to consent process | Date |

Printed name of person witnessing consent process

For IRB Use

| APPROVED by the Institutional Review Board at the University of California, Davis | |
|---|---|
| Protocol | Approved |
| 767161 | 08/20/2015 |